CLINICAL TRIAL: NCT00155389
Title: Community-based Helicobacter Pylori Eradication With Two Sequential Antibiotic Regimens for the Residents and Migrants From a High-risk Area for Gastric Cancer
Brief Title: Community-based Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 940110
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-07

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Gastric cancer; single nucleotide polymorphism
MeSH Terms: conditions — Stomach Neoplasms | interventions — Chemoprevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- H pylori eradication (Active Comparator): All enrolled subjects received chemoprevention with Helicobacter pylori eradication
  Interventions: Drug: Helicobacter pylori eradication

INTERVENTIONS:
Drug: Helicobacter pylori eradication — For subjects who received the first-line treatment, the costs included the initial 13C-UBT, one-week triple therapy (esomeprazole 40mg once daily, amoxicillin 1g twice daily, and clarithromycin 500mg twice daily), and the confirmatory 13C-UBT. For subjects in whom the initial treatment failed, the costs further included the re-treatment consisting of ten-day triple therapy (esomeprazole 40mg once daily, amoxicillin 1g twice daily, and levofloxacin 500mg once daily), and the confirmatory 13C-UBT.
  The first round of study was between 2004 and 2005, the second round was between 2008 and 2009, and the third round was between 2012 and 2013.
  Other Names: Chemoprevention

SUMMARY:
Based on a universal eradication of H. pylori in an offshore island (Matsu) with a high prevalence of gastric cancer as well as premalignant gastric lesion, we first examined the infection rate of H. pylori. Secondly, we evaluated the efficacy of clarithromycin-based triple therapy with a levofloxacin-based rescue treatment. And thirdly, we tested the hypothesis that whether the cure of H. pylori can reverse the premalignant gastric lesion. Fourth, we determine the cost-effectiveness of this intervention. The gene-environment interaction will be addressed regarding gastric cancer carcinogenesis. Finally, the incident rate of gastric cancer would be followed in this cohort.

DETAILED DESCRIPTION:
Despite the decline of global incidence, gastric cancer still affects public health substantially due to the considerable medical burden in the treatment of disease at the symptomatic stage. This fact has prompted clinicians to extend their attention from the multidisciplinary therapies to the design of preventive strategies. Gastric cancer development follows a carcinogenic process from non-atrophic gastritis, atrophic gastritis, intestinal metaplasia, dysplasia, and eventually to the adenocarcinoma. Helicobacter pylori (H. pylori) infection triggers this carcinogenic cascade and its eradication is currently the most reliable regimen to arrest the histologic progression in order to prevent gastric cancer. Emerging data have suggested that the benefit of H. pylori treatment earlier in the course of infection is larger and cannot be outweighed by a disfavored discount rate as a result of different time horizons between early treatment and later benefit of averting advanced cancer.

In the Asia-Pacific area, however, virulent strains of H. pylori infection are highly prevalent and premalignant gastric lesions may have already developed at the take-off age of active intervention. Our current knowledge remains limited in answering whether H. pylori eradication can regress these premalignant lesions and if so, what determinant can contribute to a positive response is unknown. The concept of "a point of no return" suggests that the benefit of H. pylori eradication may diminish at later stages when many types of molecular damage become irreversible. Several population-based studies, in contrast, found that the premalignant gastric lesions were potentially reversible given a sufficiently long duration free from infection. The inconsistence may reflect the facts that studies with adequate sample size and long enough follow-up are rarely available and that some important factors, such as the variation in host susceptibility to disease and dietary exposure to carcinogens, are difficult to be measured but they are likely to confound the results.

Therefore, the present study was to:

1. Determine the efficacy of a novel regimen to treat the H. pylori infection in the general population.
2. To address the question whether the premalignant gastric lesion could be reversed following the cure of infection.
3. To simulate the cost-effectiveness of this chemoprevention.
4. To use individual data to empirically calculate the cost-effectiveness of this intervention.
5. To address the host genetic susceptibility to gastric cancer development.
6. To follow-up the gastric cancer incidence following the eradication of H. pylori.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infection subjects

Exclusion Criteria:

* Prior gastrectomy; pregnant women

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2004-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Successful helicobacter eradication, change in premalignant gastric lesion, and change in gastric cancer incidence rate | 12 years

SECONDARY OUTCOMES:
Intragastric histologic change | 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Pan-Chyr Yang, PHD, Study Chair — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Lee Yi-Chia, Taipei
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Background] Lee YC, Lin JT, Wu HM, Liu TY, Yen MF, Chiu HM, Wang HP, Wu MS, Hsiu-Hsi Chen T. Cost-effectiveness analysis between primary and secondary preventive strategies for gastric cancer. Cancer Epidemiol Biomarkers Prev. 2007 May;16(5):875-85. doi: 10.1158/1055-9965.EPI-06-0758. PMID 17507609
- [Background] Liu CY, Wu CY, Lin JT, Lee YC, Yen AM, Chen TH. Multistate and multifactorial progression of gastric cancer: results from community-based mass screening for gastric cancer. J Med Screen. 2006;13 Suppl 1:S2-5. PMID 17227633
- [Background] Lee YC, Lin JT, Chen TH, Wu MS. Is eradication of Helicobacter pylori the feasible way to prevent gastric cancer? New evidence and progress, but still a long way to go. J Formos Med Assoc. 2008 Aug;107(8):591-9. doi: 10.1016/S0929-6646(08)60176-X. PMID 18678542
- [Result] Lee YC, Wu HM, Chen TH, Liu TY, Chiu HM, Chang CC, Wang HP, Wu MS, Chiang H, Wu MC, Lin JT. A community-based study of Helicobacter pylori therapy using the strategy of test, treat, retest, and re-treat initial treatment failures. Helicobacter. 2006 Oct;11(5):418-24. doi: 10.1111/j.1523-5378.2006.00432.x. PMID 16961802
- [Derived] Chiang TH, Chang WJ, Chen SL, Yen AM, Fann JC, Chiu SY, Chen YR, Chuang SL, Shieh CF, Liu CY, Chiu HM, Chiang H, Shun CT, Lin MW, Wu MS, Lin JT, Chan CC, Graham DY, Chen HH, Lee YC. Mass eradication of Helicobacter pylori to reduce gastric cancer incidence and mortality: a long-term cohort study on Matsu Islands. Gut. 2021 Feb;70(2):243-250. doi: 10.1136/gutjnl-2020-322200. Epub 2020 Aug 13. PMID 32792335
- [Derived] Lee YC, Chen TH, Chiu HM, Shun CT, Chiang H, Liu TY, Wu MS, Lin JT. The benefit of mass eradication of Helicobacter pylori infection: a community-based study of gastric cancer prevention. Gut. 2013 May;62(5):676-82. doi: 10.1136/gutjnl-2012-302240. Epub 2012 Jun 14. PMID 22698649